CLINICAL TRIAL: NCT06346444
Title: BIRS (Biomarkers in Rett Syndrome): a Long-term Observational Multicenter Study of the Natural History of Rett Syndrome to Define New Clinical and Instrumental Biomarkers
Brief Title: Biomarkers in Rett Syndrome
Acronym: BIRS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Meyer Children's Hospital IRCCS (Other); Azienda USL Toscana Nord Ovest (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Roberta Battini, Professor, IRCCS Fondazione Stella Maris
Other Study IDs: 2.780.113
Record Dates: First submitted 2024-02-22; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diagnostic test and behavioral — Questionnaires (CGI, RSBQ) and Outcome measurements (Neuroscope, EEG, Brain MRI, Bone densitometry, X-ray of thoracic and lumbosacral spine Blood biomarkers-RNA, proteins, other metabolites-)

SUMMARY:
Rett syndrome (RTT) is an X-linked genetic disorder that causes severe neurological development disorder. In its classic form, it seems to affect almost exclusively females with an incidence of up to one in 10,000 females. Patients affected by Rett Syndrome can present a wide range of symptoms, in different combinations and of varying intensity, such as slowed growth of head circumference, abnormalities in walking and balance, loss of functional use of the hands often replaced by repetitive and stereotyped hand movements like "hand washing", loss of communicative-relational skills including expressive language, epilepsy, breathing abnormalities, and osteo-muscular alterations. In light of the growing potential of clinical therapies, identification and early diagnosis are considered essential. Many disease modification strategies have been achieved through translational research studies and clinical trials that have allowed the recognition of the most effective therapeutic and clinical interventions to date.

This study arises from the need to advance in the understanding of the pathogenesis of RTT through a multicentric collaboration in order to (a) identify early biomarkers of RTT (b) delve into the alterations of interconnectivity, crucial for understanding the loss of motor functions and language through systematic collection of anamnestic, genetic, and clinical-instrumental data. The aim is to provide a valuable contribution to the study of the clinical phenotype of Rett and the identification of early interventions.

DETAILED DESCRIPTION:
The study aims to collect and analyze clinical-instrumental data from patients affected by Rett Syndrome through a prolonged monitoring program aimed at identifying disease biomarkers.

The study is a prospective observational type, with multicentric enrollment (IRCCS Stella Maris, AOU Meyer, Versilia Hospital Regional Reference Center for Rett Syndrome-USL Toscana Nord-Ovest), non-profit. New diagnosis patients and patients already included in the databases of each center will be enrolled. The cohort observational study will be completed, where possible, by a case-control study that involves the enrollment of siblings of the proband included in the study cohort.

Data regarding the registration of brain electrical activity through EEG of both the cohort and the patients' siblings, and acquisitions through Eye Tracker of the patients only, will be analyzed by Dr. Daniela Tropea's study group at Trinity College Dublin (Genetic Neuropsychiatry and Neuroscience Institute).

The study is expected to start immediately after the approval of the protocol by this Ethics Committee.

The study is expected to last four years. The study involves the enrollment of every case of Rett syndrome in the developmental age attending one of the Italian centers and an annual follow-up with clinical and instrumental controls provided by a dedicated path.

Sample Size The sample size has been estimated according to the syndrome's prevalence in the general population and based on the number of retrospective patient samples affected by Rett Syndrome.

The study plans to enroll approximately 100 patients consecutively, according to a pre-established schedule that includes observations and evaluations provided by the protocol.

FOLLOW-UP PROCEDURE The follow-up of each patient will be carried out annually through clinical monitoring and instrumental application of what is listed in the primary endpoint except for the brain MRI, whose repetition if necessary will be agreed upon based on the evolution of the clinical picture.

DEFINITION OF STUDY CONCLUSION The end of the monitoring of patients is expected upon reaching the age of 18 years.

DATA MANAGEMENT For each recruited patient, after deliberation through informed consent, data contained within the clinical record will be collected. At recruitment, data related to diagnosis, gestational age at birth, auxological parameters at birth, Apgar score, main clinical anamnestic data related to the perinatal period, and outcome of neuroimaging assessments carried out (for example, brain MRI, transfontanellar cerebral ultrasound) will be acquired and recorded in a specific database.

To protect privacy, each patient will be assigned a numeric code, therefore the database will not contain any demographic data, and access will be protected by a password and limited to personnel involved in the study only. The database will be progressively implemented with the outcomes of the assessments, acquired systematically, according to the correspondence code of the individual subject. The EEG video recording data will be accessible from the clinical documentation and coded systematically. The EEG data and the acquisitions through Eye Tracker obtained in the Italian enrollment centers will be analyzed at Trinity College Dublin in an anonymous manner through identification by numeric code and only after signed consent from the parents.

DATA CONSERVATION The data managers and the measures of anonymization will be the responsibility of the main experimenters of the study. All data will be stored in secure places and on password-protected files, at the patient's home institute.

ETHICAL CONSIDERATIONS The study conforms to the ethical principles recognized for clinical experimentation, to the principles of good clinical practice.

The protocol has been submitted for approval to the ethical committee and/or competent authority.

ACQUISITION OF INFORMED CONSENT AND DATA PROCESSING At the time of the direct interview with the families, a detailed explanation will be provided orally and a written informative note (which will remain with the parents). The importance of the study and the data used for the purposes of our study will also be explained, specifying the request for release for the compilation of the database, however under an identification code.

The paper documents related to informed consent will be handed over to the family so that they can be read and understood in their entirety and retrieved following a subsequent interview in which the parents can ask clarifying questions and definitively confirm their consent to the study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects aged between 0 and 18 years with Rett Syndrome, classic (mutation of the MECP2 gene) and Rett variants (CDKL5, FOXG1 mutations, and other MECP2 mutations), genetically confirmed:

  * newly diagnosed
  * previously diagnosed if possessing data recorded and stored in the enrollment centers' records;
  * upon written informed consent from the parents.
* Siblings of the probands of any age who will undergo EEG registration will also be enrolled.

Exclusion Criteria:

• Patients with Rett Syndrome presenting a compromise in the general health status to such an extent that it makes it impossible to apply the clinical-instrumental evaluation and monitoring tools used for the study.

Ages: 0 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample size has been estimated according to the syndrome's prevalence in the general population and based on the number of retrospective patient samples affected by Rett Syndrome and Reti-like Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Age at diagnosis | every year for four years
Mutation in MECP2 | every year for four years
  Number of different single variant
Neuroscope alterations | every year for four years
  NeuroScope is an advanced viewer for neurophysiological and behavioral data: it can display local field potentials (LFPs), neuronal spikes and behavioral events.
Electroencephalogram (EEG) alterations | every year for four years
Brain magnetic resonance imaging (MRI) alteration | every year for four years
Bone densitometry alterations | every year for four years
Thoracic radiographic alterations | every year for four years
Lumbosacral spine radiographic alterations | every year for four years
Clinical Global Impression (CGI) scale | every year for four years
  The CGI scale has two components-the CGI-Severity, which rates illness severity of ill (Score from 1 to 7, where 1 is normal and 7 severely ill) , and the CGI-Improvement, which rates change from the initiation (baseline) of observation (Score from 1 to 7, where 1 is very much improved since the initiation of observation and 7 is very much worse since the initiation of observation)
The Rett Syndrome Behavioural Questionnaire (RSBQ) | every year for four years
  The Rett Syndrome Behaviour Questionnaire (RSBQ) assesses the severity of neurobehavioral problems from the perspective of the caregiver. The RSBQ consists of 45 items of which 38 items are grouped into 8 domains/subscales that reflect the core features (General Mood; Breathing Problems; Hand Behaviors; Repetitive Face Movements; Body Rocking and Expressionless Face; Nighttime Behaviors; Fear/Anxiety; and Walking/Standing) and 7 items are grouped into a subscales classed as "uncategorized" but contribute to the overall total score. Each item is rated on a Likert scale as 0 (behavior "not true"), 1 (behavior "somewhat or sometimes true") or 2 (behavior "often true"), with the total score ranging from 0 to 90 (higher scores indicate increased severity)

SECONDARY OUTCOMES:
Alterations of neurovisual functions | every year for four years
Possibility of applying alternative forms of communication to verbal communication | every year for four years
  Possibility of applying alternative forms of communication to verbal communication (in patients presenting with the absence of expressive language) through the application of the EYE TRACKER device (Tobii Dyanvox) that uses near-infrared lighting in combination with high-definition cameras to project light into the eye and record the direction reflected by the cornea

CONTACTS AND LOCATIONS:
Locations (4):
- Trinity College Institute of Neuroscience, Lloyd Building, D2, Dublin, Ireland
- Italy (3):
  - Ospedale Versilia Centro di Riferimento, Lido di Camaiore, Lucca
  - IRCCS Fondazione Stella Maris, Calambrone, Pisa
  - AOU Meyer, Florence

IPD SHARING:
Plan to Share IPD: No